CLINICAL TRIAL: NCT02391168
Title: A Multi-center, Prospective Cohort Study on the Natural History of Fatty Liver Disease in China
Brief Title: Fatty Liver Disease Collaborative Research in China
Acronym: FLDCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fatty Liver and Alcoholic Liver Disease Study Group, China (Other)
Collaborators: Unimed Scientific Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FLD2015
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Fatty Liver; Fatty Liver, Alcoholic; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Fatty Liver; Fatty Liver, Alcoholic; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Liver tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
A multi-center, prospective cohort study on the natural history of fatty liver disease in China

DETAILED DESCRIPTION:
This is a multicenter, prospective and open-enrollment epidemiologic study. All the patients with liver biopsy-proven macrovesicular steatosis (>5%) will be enrolled in the baseline cross-sectional analysis. Those who are either diagnosed as NAFLD or ALD, if meeting all the inclusion and exclusion criteria, will be enrolled in the following cohort study, will be followed up after 1 year, 3 years and 5 years with a visit window of +1 month.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed fatty liver disease, confirmed by liver biopsy.
* Specific biopsy requirements: qualified biopsy specimen within 6 months, >5% hepatocytes show macrovesicular steatosis under HE staining and X10 microscope.
* Only patients with NAFLD or ALD are eligible for the 5-year follow-up cohort study.
* Willing to participate in the long-term follow-up and cooperative.
* Able to provide informed consent file.

Exclusion Criteria:

* Unable to provide informed consent.
* Patients are eligible for baseline cross-sectional analysis but not eligible for the cohort section, if having any of the following condition:

  1. Any end-stage liver disease.
  2. Any malignant tumor.
  3. Any infection of hepatitis virus or HIV.
  4. Any congenital liver disease such as Wilson disease.
  5. Any other serious disease of projected survival < 5 years.
  6. Combined NAFLD and ALD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any person with fatty liver disease
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
liver cirrhosis | 5 years

SECONDARY OUTCOMES:
liver cancer | 5 years
liver failure | 5 years
type 2 diabetes | 5 years
cardiovascular and cerebrovascular events | 5 years
death | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiangao Fan, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (6):
- China (6):
  - Zhangzhou Zhengxing Hospital, Zhangzhou, Fujian
  - Shandong Provincial Hospital, Ji'nan, Shandong
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - Shanghai Xinhua Hospital, Shanghai